CLINICAL TRIAL: NCT06247592
Title: Comparison of Greater Occipital Nerve Block and Pulse Radiofrequency in Patients With Chronic Migraine
Brief Title: Pulse Radiofrequency and Occipital Nerve Block for Chronic Migraine Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Esra Ertilav, Assoc.Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023/03
Record Dates: First submitted 2024-01-05; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Chronic Migraine, Headache; Block; Occipital Neuralgia
Keywords: chronic migraine; greater occipital nerve block; pulse radio frequency; pain management
MeSH Terms: conditions — Headache; Bites and Stings; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency group (Experimental): Pulse radiofrequency will be applied at 42 degrees for 240 seconds with a channel placed near the greater occipital nerve.
  Interventions: Procedure: Greater occipital nerve pulse radiofrequency
- Block group (Active Comparator): Nerve blockade will be applied to the greater occipital nerve with 5 cc 2% prilocaine.
  Interventions: Procedure: Greater occipital nerve block

INTERVENTIONS:
Procedure: Greater occipital nerve block — Pulse Radiofrequency application to the greater occipital nerve will be applicated after radiofrequency cannula placed near the greater occipital nerve location at 42 degree, for 240 seconds.
  Arms: Block group
Procedure: Greater occipital nerve pulse radiofrequency — The greater occipital nerve will be blocked with 5 cc 2% prilocaine.
  Arms: Radiofrequency group

SUMMARY:
In this study, the effect of nerve blockade and radiofrequency treatment applied to the nerve on pain in chronic migraine patients will be investigated.

Occipital nerve blockade group (control group): Depending on the location of the pain, blockade will be applied unilaterally or bilaterally with 5 cc of 2% prilocaine for each sıde.

Pulse Radiofrequency application to the greater occipital nerve will be applicated after radiofrequency cannula placed near the greater occipital nerve location with 42 degree, for 240 seconds.

DETAILED DESCRIPTION:
Patients between the ages of 18-60 years, who were resistant to medical treatment and diagnosed with chronic migraine according to ICHD-3 beta criteria (migraine pain for more than 15 days in the last 3 months) who applied to the Neurology and Algology outpatient clinic were included in the study.

All procedures were performed with the patient in the prone position, using anatomical landmarks in the target areas. For Gon Blockade, the target point for the greater occipital nerve was identified along a line connecting the external occipital protuberance to the mastoid process (usually 1.5-3 cm lateral to the midline) and one-third of the distance medial to the artery at the level of the superior nuchal process. After local anesthesia with skin-subcutaneous 1% lidocaine, bone contact was obtained using a 25-gauge needle. For Pulse Radiofrequency, the target point for the greater occipital nerve was determined as one third of the distance medial to the artery along a line connecting the external occipital protuberance to the mastoid process (usually 1.5-3 cm lateral to the midline) and at the level of the superior nuchal process. After local anesthesia with skin-subcutaneous 1% lidocaine, a 5 cm long 20 gauge radiofrequency needle with a 5 mm active tip was inserted close to the targeted nerve. Sensory and motor electrical stimulation was performed to elicit a compatible paresthesia response in the occipital distribution. Pulsed radiofrequency was applied at 42 degrees C for 240 seconds. Patients were observed after the procedure. Patients were observed before and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-60 years of age diagnosed with chronic migraine according to IHS criteria

Exclusion Criteria:

* Pregnancy
* Major psychiatric disorder
* Bleeding diathesis
* Local infection
* Allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Pain Relief | 1 and 3 months
  Compare the efficacy of blockade procedure applied to the greater occipital nerve with pulse radiofrequency therapy in terms of pain relief with Visual Analog Scale in chronic migraine patients.The visual analog scale (VAS) is numbered from 0 to 10. 10 is the most severe pain 0: no pain at all

SECONDARY OUTCOMES:
Disability, Quality of life | 1 and 3 months
  Compare the efficacy of occipital nerve block with pulse radiofrequency therapy in terms of disability and quality of life with MIDAS (Migraine Disability Assessment) questionnaire win chronic migraine patients. The MIDAS classification is numbered from 0 to 4. 4 means severe disability 0: no disability at all

CONTACTS AND LOCATIONS:
Overall Officials: Esra Ertilav, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Esra Ertilav, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
YES